CLINICAL TRIAL: NCT05945836
Title: Excess Cement and Peri-implant Disease: A Cross-sectional Clinical Endoscopic Study
Brief Title: Peri-implant Disease and Prosthetic Cement: Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Marco Montevecchi, Assistant professor, University of Bologna
Other Study IDs: peri-implant/cement
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis
Keywords: Dental implants; Peri-implant diseases; Excess cement; Implant prosthesis; Endoscopy
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the present clinical study project, of a cross-sectional observational nature, is to evaluate the presence of submucosal cement residues through endoscopic visualization in clinical situations with peri-implant disease.

The secondary objective is to investigate the potential correlation between the severity of the pathological condition and the spatial position of cement residues in relation to the implant-prosthetic unit.

For each subject, the following data were collected: gender, age, periodontal history, smoking habits, reasons for implant rehabilitation (trauma, caries, periodontitis, agenesis, other), the position of the implant in the oral cavity, elapsed time between prosthetic rehabilitation and pathological condition. If the deposit was recognized as cement residue, its presence was recorded, and the anatomical position of the cement residue (mesial, distal, lingual/palatal, vestibular) and the spatial position of cement residues in relation to the implant-prosthetic unit were collected.

ELIGIBILITY:
Inclusion Criteria:

* at least one single-implant with cemented restoration and clinical-radiographic signs of peri-implant disease
* patients with previous periodontitis had to have a healthy but reduced periodontium

Exclusion Criteria:

* neuromotor pathologies or morphological-dysfunctional alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutively, all subjects over 18 years of age presenting at least one cemented single-implant restoration with clinical and radiographic signs of peri-implant disease were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of submucosal cement | The analysis was conducted during the endoscopic examination between October 29, 2018, and July 19, 2019.
  A clinical examination of the submarginal implant area was performed using endoscopic techniques (DV2, Dental View, Irvine, CA). The analysis was conducted in an atraumatic manner, and local anesthesia infiltration (2% Mepivacaine with 1:100,000 adrenaline) was administered only upon patient request. During the endoscopic investigation, once a deposit was identified, its consistency and adhesion were assessed using water irrigation or, less frequently, a probe. Only for solid deposits, a differential analysis between calculus and cementum was conducted. Cementum was identified by its characteristic white reflectivity, in contrast to subgingival calculus, which appeared yellow or brown, depending on the intensity and distance of the incident light beam.

SECONDARY OUTCOMES:
Spatial position of submucosal cement | The analysis was conducted during the endoscopic examination between October 29, 2018, and July 19, 2019.
  If the deposit was recognized as cement residue, its presence was recorded, and the following clinical data were collected:
  * Distance between mucosal margin and prosthetic closure margin at the site of the cement residue: MM-PM = Mucosal Margin - Prosthetic Margin
  * Distance between prosthetic closure margin and implant platform at the site of the cement residue: PM-IP = Prosthetic Margin - Implant Platform
  * Distance between the most apical portion of the cement residue and implant platform: AC-IP = Apical Cement - Implant Platform

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montevecchi, DDS, Study Chair — Alma Mater Studiorum - University of Bologna
Locations (1):
- Alma Mater Studiorum - University of Bologna, Department of Biomedical and Neuromotor Sciences, School of Dentistry - Division of Periodontology and Implantology., Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available when the research will be published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available when the research will be published
Access Criteria: On request to the main investigator